CLINICAL TRIAL: NCT00253227
Title: Galantamine in the Treatment of Alzheimer's Disease: Flexible Dose Range Trial
Brief Title: A Study of the Safety and Effectiveness of a Flexible Dose of Galantamine Versus Placebo in the Treatment of Patients With Alzheimer's Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR006028
Record Dates: First submitted 2005-11-10; First posted 2005-11-15 (Estimated); Last update posted 2011-05-18 (Estimated); Status verified 2010-11

CONDITIONS: Alzheimer Disease; Dementia
Keywords: Alzheimer's disease; dementia; brain disease; memory loss; galantamine; placebo
MeSH Terms: conditions — Alzheimer Disease; Dementia; Brain Diseases; Memory Disorders | interventions — Galantamine

INTERVENTIONS:
Drug: galantamine hydrobromide

SUMMARY:
The purpose of this study is to evaluate the safety and effectiveness of galantamine (a drug for treating dementia) versus placebo in the treatment of patients with Alzheimer's disease using a flexible dose design.

DETAILED DESCRIPTION:
Dementia is a chronic, progressive brain disease that may involve a number of symptoms, including memory loss and changes in personality, behavior, judgment, attention span, language and thought. The most common type of dementia is Alzheimer's disease. Over time, patients with Alzheimer's disease may lose ability to perform daily tasks related to personal care (for example bathing, dressing, eating) and may be unable to handle money or travel to familiar places. Several small clinical trials have shown galantamine to be safe and effective in treating the symptoms associated with Alzheimer's disease. Doses studied have ranged from 22.5 - 45 mg/day, with galantamine administered two or three times daily. Additional information is needed to determine the optimal dose regimen for galantamine in the treatment of Alzheimer's' disease. This multicenter, double-blind, placebo-controlled (neither the patient nor the study doctor know the dose of galantamine being given) study evaluates the safety and effectiveness of galantamine in the treatment of patients with Alzheimer's disease using a flexible dose regimen of two doses of galantamine. The flexible dose regimen was chosen in order to allow the physicians to give each patient an optimal dose of galantamine, to simulate what might be done in clinical practice, rather than to require all patients to receive a fixed dose throughout the study. All patients initially receive placebo for a 1-month period and then receive one of two doses of galantamine (beginning with 4 mg twice daily and gradually increasing to 12 or 16 mg twice daily) or placebo for 3 months. The primary measures of effectiveness include the change from baseline to the end of treatment in the ADAS-cog/11 score (Alzheimer's Disease Assessment Scale: sum of 11 cognitive items) and the CIBIC-plus score (Clinician's Interview Based Impression of Change - Plus Caregiver Input). Additional measures of effectiveness assessed at the end of the treatment include the ADAS-cog/13 score (Alzheimer's Disease Assessment Scale: sum of 13 cognitive items), the Disability Assessment for Dementia (DAD) score and the Neuropsychiatric Inventory (NPI)) score. Safety evaluations (incidence of adverse events, quality of sleep (using the Pittsburgh Sleep Scale), electrocardiograms (ECGs), physical examinations, laboratory tests) are performed throughout the study. Blood samples are taken throughout the study to determine the concentration of drug in the blood. Patients who complete this study will have the option to receive open-label galantamine in a separate study. The study hypothesis is that galantamine administered in either dose is effective in the treatment of Alzheimer's disease as compared with placebo and well tolerated, and that using a flexible dose regimen will allow these patients to receive an individualized dose of galantamine that is effective and well tolerated. Galantamine tablets (or placebo), 12 or 16 mg by mouth twice daily for 3 months, beginning with 4 mg twice daily and gradually increasing to 12 or 16 mg twice daily.

ELIGIBILITY:
Inclusion Criteria:

* Outpatients with a diagnosis of Alzheimer's disease according to the National Institute of Neurological and Communicative Disorders and the Alzheimer's Disease and Related Disorders Association (NINCDS-ADRDA) criteria (including patients living independently in residential homes for the elderly or day patients)
* have mild to moderate dementia, as evidenced by a, Mini-Mental Status Examination (MMSE) score of 11 - 24, and a score of at least 12 on the cognitive portion of the Alzheimer's Disease Assessment scale (ADAS-cog)
* history of at least 6 months of gradual and progressive cognitive decline
* have a consistent informant to accompany the patient on scheduled visits

Exclusion Criteria:

* Neurogenerative disorders such as Parkinson's disease
* dementia caused by small strokes or cerebrovascular disease
* cognitive impairment resulting from acute cerebral trauma, cerebral damage due to a lack of oxygen, vitamin deficiency, infections such as meningitis or AIDS, significant endocrine or metabolic disease, mental retardation or a brain tumor
* having epilepsy, significant psychiatric disease, active peptic ulcer, clinically significant liver, kidney or lung disorders or heart disease
* Females of child bearing potential without adequate contraception

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 387 (Actual)
Dates: Start 1997-07; Study Completion 1998-12 (Actual)

PRIMARY OUTCOMES:
Change from baseline to the end of treatment in ADAS-cog/11 (Alzheimer's Disease Assessment Scale: sum of 11 cognitive items) and CIBIC-plus (Clinician's Interview Based Impression of Change - Plus Caregiver Input) scores

SECONDARY OUTCOMES:
Change from baseline in ADAS-cog/13, DAD and NPI scores to the end of treatment; Incidence of adverse events; Pittsburgh Sleep Scale score; Changes in laboratory tests, ECGs and physical examinations

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.

REFERENCES:
- [Result] Rockwood K, Mintzer J, Truyen L, Wessel T, Wilkinson D. Effects of a flexible galantamine dose in Alzheimer's disease: a randomised, controlled trial. J Neurol Neurosurg Psychiatry. 2001 Nov;71(5):589-95. doi: 10.1136/jnnp.71.5.589. PMID 11606667
- [Derived] Lim AWY, Schneider L, Loy C. Galantamine for dementia due to Alzheimer's disease and mild cognitive impairment. Cochrane Database Syst Rev. 2024 Nov 5;11(11):CD001747. doi: 10.1002/14651858.CD001747.pub4. PMID 39498781
- See also: A study of the safety and effectiveness of a flexible dose of galantamine in patients with Alzheimer's disease — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=700&filename=CR006028_CSR.pdf